CLINICAL TRIAL: NCT05753410
Title: Feasibility and Acceptability of an App-Based Mindfulness Training for Individuals With Anorexia Nervosa and Bulimia Nervosa
Brief Title: App-Based Mindfulness Training for Individuals With Anorexia Nervosa and Bulimia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeshiva University (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Margaret Sala, Assistant Professor, Yeshiva University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20204635
Record Dates: First submitted 2023-02-21; First posted 2023-03-03 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa; Anorexia Nervosa, Atypical; Bulimia; Atypical
Keywords: Anorexia Nervosa; Bulimia Nervosa; Mindfulness Training; Digital Intervention
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa; Bulimia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful Courage (Experimental): Mindful Courage is a digital intervention including mindfulness and cognitive behavioral elements for individuals with anorexia nervosa or bulimia nervosa. Mindful Courage will consist of 8-weeks of self-guided modules which will be completed over the course of 8 weeks. Elements included in the intervention include psychoeducation, self-monitoring, regular eating, body image, values clarification, and mindful awareness and acceptance. Participants learn a range mindfulness skills and practice a range of mindfulness meditations. Participants will also receive phone coaching. Homework consists of meditation practices.
  Interventions: Behavioral: Mindful Courage

INTERVENTIONS:
Behavioral: Mindful Courage — Self-guided online intervention

SUMMARY:
We will evaluate the acceptability and feasibility of a 8-week long digital mindfulness-based intervention for anorexia nervosa and bulimia nervosa.

This study is a prospective single-arm trial during the intervention development phase. Following this phase, after the intervention has been further developed, a subsequent study (with a different clinicaltrials.gov identification #) will utilize a randomized control trial design.

DETAILED DESCRIPTION:
Procedures include completing: (1) pre-intervention screening assessment; (2) brief daily assessments for the first and last weeks of the study (4 times per day); (3) an initial baseline visit; (4) 8-week web-based intervention (3) a post-intervention assessment (8-weeks after baseline); and (4) a brief 8-week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Can read and write in English
* Meet diagnostic DSM 5 diagnostic criteria for anorexia nervosa, bulimia nervosa, or atypical anorexia nervosa/bulimia nervosa
* Owns a smartphone
* Willing and able to participate in an eight-week long research study
* Have a private quiet space at home or headphones to complete modules
* Completed one month or more of eating disorder treatment
* Currently enrolled in eating disorder treatment

Exclusion Criteria:

* Fail to meet above-listed inclusion criteria
* Current alcohol or drug dependence
* Current untreated psychotic or bipolar disorder
* Current suicidal intent
* Significant cognitive impairment that would impair the ability to use Mindful Courage effectively
* BMI <15 or medically unstable
* Currently receiving residential/inpatient treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Feasibility | 8-week treatment period
  Module completion, ranging from 0 to 100%
Acceptability dimensions | 8-week treatment period
  Single-items measuring ratings of acceptability dimensions, including usability, understandability, engage-ability, visual appeal, helpfulness, skill acquisition, and confidence implementing skills ratings. Scores for each item range from 1 to 5, , with higher scores indicating better acceptability.

SECONDARY OUTCOMES:
Change in Eating Disorder Symptoms | Baseline to post-treatment (8-weeks) and through 2-month follow-up
  Eating Disorder Examination-Questionnaire (EDE-Q). Total scores are the average of each of the subscales, and range from 0 to 6. Higher scores indicate higher eating disorder symptoms.
Change in Emotion Dysregulation | Baseline to post-treatment (8-weeks) and through 2-month follow-up
  Difficulties in Emotion Regulation Short Form (DERS-SF). Total scores are the average of each of the subscales, and range from 1 to 5. Higher scores indicate more emotion dysregulation
Change in Body Dissatisfaction | Baseline to post-treatment (8-weeks) and through 2-month follow-up
  Body Shape Questionnaire (BSQ). Total scores are the total across the items, and range from 34 to 204. Higher scores indicate greater body dissatisfaction.
Savoring Beliefs | Baseline to post-treatment(8-weeks) and through 2-month follow-up
  Savoring Beliefs Inventory (SBI). Total scores are the total across the positively-anchored and negatively-anchored items, and could range from -72 to 72. Higher scores reflect stronger endorsement of savoring beliefs.
Psychosocial Impairment | Baseline to post-treatment (8-weeks) and through 2-month follow-up
  Clinical Impairment Assessment Questionnaire (CIA). Total scores are the total of the items, and range from 0 to 48. Higher scores indicate greater psychosocial impairment associated with an eating disorder.
Change in Mindfulness | Baseline to post-treatment (8-weeks) and through 2-month follow-up
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R). Total scores range from 0 to 40, with higher scores indicating greater mindfulness.

CONTACTS AND LOCATIONS:
Locations (1):
- Margaret Sala, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided